CLINICAL TRIAL: NCT01384942
Title: The Development and Pilot Testing of Meaning-based Group Counselling Intervention for Bereavement
Brief Title: Meaning-based Group Counselling for Bereavement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Christopher J. MacKinnon, Psychologist, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 002645; NCT01285128 (obsolete NCT alias)
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-08

CONDITIONS: Grief; Bereavement
Keywords: Bereavement; Grief; Mourning; Loss; Death; Meaning; Group; Counseling; Psychotherapy; Uncomplicated; Support
MeSH Terms: conditions — Death

ARMS (2):
- Meaning-Based Bereavement Group (Experimental)
  Interventions: Behavioral: Meaning-Based Bereavement Group
- Conventional Bereavement Group (Active Comparator)
  Interventions: Behavioral: Conventional Bereavement Group

INTERVENTIONS:
Behavioral: Meaning-Based Bereavement Group — A 12 week bereavement counselling group with tasks and themes that focus on re-constructing meaning following death.
  Arms: Meaning-Based Bereavement Group
Behavioral: Conventional Bereavement Group — An 8 week traditional bereavement group that follows a more conventional approach to grief support.
  Arms: Conventional Bereavement Group

SUMMARY:
Given that individuals in bereavement tend to experience substantial psychological distress in the first two years following loss, individuals seeking psychological support will need appropriate services grounded in sound empirical scholarship. There is a lack of studies assessing bereavement groups, despite groups being one of the most common forms by which such services are offered. The prominent and emerging process of meaning-reconstruction in bereavement research is theorized to lead to better psychological adjustment and prevent more prolonged grief reactions. The principal objective of this study is to compare two types of group counseling for individuals in bereavement: A novel meaning-based bereavement counseling group and a conventional bereavement support group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting for bereavement services that have experienced a death-related loss within 6 weeks to 2 years of the first meeting of the group, and are experiencing an uncomplicated grief response will be invited to participate.
* Individuals will be assessed for their ability to participate in a group counselling context as well as an uncomplicated grief trajectory. Participants must be 18 years of age or older, have sufficient ability to communicate in English, as well as read English.

Exclusion Criteria:

* Following a clinical/diagnostic interview and administration of the PG-13 (Prolonged Grief Disorder-13, Prigerson et al., 2009), individuals experiencing a complicated/prolonged grief trajectory are excluded.
* Furthermore, individuals whose cognitive condition might make the study burdensome or impossible for them are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Grief | 24 weeks
  Descriptive statistical analysis (e.g., means, standard deviations, percentage of scale range improvements) will be conducted on the pre-test, post-test, and follow-up scores for both the experimental and control group on the following outcome measures
  (1) Grief: Revised Grief Experience Inventory; Core Bereavement; Hogan Grief Reaction Checklist
Meaning | 24 weeks
  Descriptive statistical analysis (e.g., means, standard deviations, percentage of scale range improvements) will be conducted on the pre-test, post-test, and follow-up scores for both the experimental and control group on the following outcome measures
  (1) Meaning: Purpose in Life Test; The Grief and Meaning-Reconstruction Inventory; The Integration of Stressful Life Experiences Scale
Depression | 24 Weeks
  Descriptive statistical analysis (e.g., means, standard deviations, percentage of scale range improvements) will be conducted on the pre-test, post-test, and follow-up scores for both the experimental and control group on the following outcome measures
  (1) Depression: Center for Epidemiologic Studies Depression Scale
Anxiety | 24 Weeks
  Descriptive statistical analysis (e.g., means, standard deviations, percentage of scale range improvements) will be conducted on the pre-test, post-test, and follow-up scores for both the experimental and control group on the following outcome measures
  (1)Anxiety: State-Trait Anxiety Scale

CONTACTS AND LOCATIONS:
Locations (1):
- S.M.B.D. Jewish General Hospital / Hope and Cope Program, Montreal, Quebec, Canada